CLINICAL TRIAL: NCT06724497
Title: Evaluating the Accuracy of Soft Tissue Prediction in Patients With Mandibular Prognathism After Orthognathic Surgery Using Handheld Scanner Versus Optical Scanner A Prospective Clinical Trial
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Fahim, PhD candidate, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 337
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Mandibular Prognathism; Orthognathic Surgery
Keywords: Prognathism; soft tissue prediction; face scanner; handheld scanner; optical scanner; orthognathic surgery; prediction accuracy
MeSH Terms: conditions — Malocclusion, Angle Class III; Prognathism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with mandibular prognathism (Other): same patient will be scanned twice using both devices the optical face scanner and the handheld optical scanner
  Interventions: Procedure: face scanning pre and post orthognathic surgery

INTERVENTIONS:
Procedure: face scanning pre and post orthognathic surgery — patient will be scanned pre operative using both scanners and then undergo orthognathic surgery then will be rescanned again 6 montsh later

SUMMARY:
Aim of study: To evaluate the accuracy of soft tissue prediction in orthognathic surgery using handheld scanners versus optical scanners.

Research hypothesis (null hypothesis): there is no difference in prediction accuracy between laser scans and handheld scans.

Primary objective: To evaluate The Accuracy of soft tissue prediction in orthognathic surgery using handheld scanner versus laser scanner

.

Secondary objective:

To evaluate scanning time, cost efficiency, and ease of use. patients will be treated from mandibular prognathism using only mandibular set back or bimaxillary surgery After six months postoperatively, 3D facial scans is obtained and exported to software to perform superimposition of the predicted and post operative results to assess the accuracy of soft tissue prediction By measuring the difference in millimeter between prespecified points

DETAILED DESCRIPTION:
Aim of study: To evaluate The Accuracy of soft tissue prediction in orthognathic surgery using handheld scanner versus optical scanner.

Research hypothesis (null hypothesis) that there is no difference in prediction accuracy between laser scans and handheld scans.

Primary objective: To evaluate The Accuracy of soft tissue prediction in orthognathic surgery using handheld scanner versus laser scanner .

Secondary objective:

To evaluate scanning time, cost efficiency, ease of use. 8. Trial design

One group of patients will be assigned to this trial:

One group: same patient will be scanned by both devices preoperatively and post operatively.

Trial design: prospective clinical trial( diagnostic accuracy study )

III. Methods A) Participants, interventions & outcomes 9. Study settings: Oral and Maxillofacial Surgery clinic, Faculty of Dentistry, Cairo University. 10. Eligibility criteria:

Inclusion criteria:

* Patients with facial mandibular prognathism that requires orthognathic surgery.
* Age (18- 50years).
* Patients are willing for the surgical procedure and follow-up, with informed consent (appendix 1).

Exclusion criteria:

* Dental malocclusion that could be treated with orthodontic treatment only.
* Patients with contraindications for general anesthesia.
* Patient on radiotherapy.
* Patients suffer from bone disease. 11. Interventions Preoperative Investigations
* From the point of eligibility for general anesthesia, complete blood picture, body weight, urine albumin, blood glucose level, kidney and liver function.
* Administration of peri-operative antibiotics.
* A multi-slice CT scan will be demanded in a form of DICOM files ( Digital Imaging and Communications in Medicine) for proper diagnosis and confirmation of patient compatibility to the eligibility criteria and digital planning of the study group.
* For each patient soft tissue scanning will be taken using cr-scan ferret scanner (Creality,shinzen,china) file will be imported to specialized software PROPLAN CMF™ (Leuven, Belgium)
* then soft tissue scan will be done using optical scanner then the file will be imported to a specialized software PROPLAN CMF™ (Leuven, Belgium)
* for segmentation process and superimposition of the soft tissue scan and the CT dicom file and planning the osteotome and fabrication of surgical guide for accurate positioning and fixation of bone segment.
* Sterilization of the patient-specific plates and splints
* For hemostasis an Epinephrine solution in dilution of 1:200.000 with lignocaine 0.5 mg\ml injected along lines of surgical incisions 5 min before the surgery.

The surgical technique:

All surgeries will be carried out with endotracheal intubation under general anaesthesia.

1. the planned osteotomies are performed on the upper jaw (maxilla), lower jaw (mandible), or both, depending on the treatment plan.
2. Repositioning of Jaw Bones: into the planned alignment to correct the underlying skeletal discrepancies. This may involve moving the jaws forward, backward, upward, or downward as needed to achieve proper facial harmony and function.
3. Stabilization: using plates and screws to stabilize the bones in their new position. This promotes proper healing and ensures long-term stability of the surgical outcome.

Postoperative Management:

* Postoperative instructions include a sleeping in a supine position semi-up righted, Strict oral hygiene measures.
* Postoperative medications include prophylactic broad-spectrum antibiotics for 5 days' post operatively, nonsteroidal anti-inflammatory drug, diclofenac.

Suture will be removed after 7 days post operative.

Accuracy measurement:

After six months post operative 3d facial scans is obtained and exported to software to perform superimposition of the predicted and post operative results to assess the accuracy of soft tissue prediction By measuring the difference in millimeter between prespecified points

1-full face 2-subnasal 3-labrale superioris 4- labrale inferioris 5-pogonion 6- corners of the mouth Then the degree of accuracy will be measured in percentage

Follow up:

All patients will undergo CT scans before the first follow-up 3 days postoperative.

Strategies to improve adherence to intervention protocol:

* The patient will be educated about the treatment protocol including a rationale for each step and an emphasis on the significance of follow-up appointments and home. Medicine.
* All patients will be given reminder phone calls at the time of the predetermined follow updates.

Criteria for discounting allocated intervention Uncooperative patients are refusing treatment and follow up.

Side effects and the degree of risk and expected to occur and how to deal with them Any temporary or permanent adverse effect will be recorded, documented, and treated including (facial asymmetry, pain trismus, paranesthesia, edema, and infection, flap dehiscence and plate exposure).

In the event of temporary side effects such as swelling or numbness, the patient will be followed up periodically and the necessary medications will be prescribed to get rid of these symptoms.

If facial asymmetry occurs after the operation, the necessary corrective measures will be taken, such as following up with the orthodontist or repeating the surgical procedure if necessary.

the event of a bacterial infection, the patient will be given the necessary medications after examination and confirmation of the source and cause of the infection and plate removal if needed

For patients equal to and less than 21 years old, a written consent should be obtained from their parents or guardian that they understand the treatment plan and agree for their children to undergo the surgical procedure and they understand the harms and side effects of this procedure and they will adhere to the follow up plans.

12. Outcomes:

Outcome name Measuring Device Measuring Unit Primary

Soft tissue prediction accuracy

Computer Software Difference between prespecified measuring points in mm 1-full face 2-subnasal 3-labrale superioris 4- labrale inferioris 5-pogonion 6-corners of the mouth

Then turned into percentage Secondary scanning time Stopwatch seconds

Ease of use

scale Score from 1-10

1 very easy 10 very hard Cost efficiency Cost price pounds

* For standardization of follow up the accuracy of soft tissue prediction will be measured by superimposition the planning with the postoperative 3D scan of the patient Then, the distance between the planning and the scan will be estimated in millimeters. Then software will give a percentage
* scanning time will be estimated in seconds.
* Ease of use
* cost 13. Participant timeline Patient will be treated in (5) visits . Visit 1: case evaluation and diagnosis, request CT scan and soft tissue scan. Visit 2: patient education, anesthesiologist consultation, consent signing. Visit 3: operation day. Visit 4: one week after surgery clinically evaluation and Patient questionnaire will be filled .

Visit 5: six months postoperative clinical follow up and post operative soft tissue scanning.

Time Procedure Visit 1 Day 0 Case evaluation and diagnosis, request CT scan and soft tissue scan.

Visit 2 Week 1 Patient education, consent signing, anesthesiologist consultation.

Visit 3 Week 2 Surgical procedure. Visit 4 Week 3 First follow up, questionnaire,

Visit 5 Week 26 postoperative CT scan evaluation and soft tissue scanning and suture removal.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with facial mandibular prognathism that requires orthognathic surgery.

  * Age (18- 50 years).
  * Patients are willing for the surgical procedure and follow-up, with informed consent

Exclusion Criteria:

* • Dental malocclusion that could be treated with orthodontic treatment only.

  * Patients with contraindications for general anesthesia.
  * Patient on radiotherapy.
  * Patients suffer from bone disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-09-24 (Estimated)

PRIMARY OUTCOMES:
soft tissue prediction accurace | six months after surgery
  3d facial scans is obtained and exported to software to perform superimposition of the predicted and post operative results to assess the accuracy of soft tissue prediction By measuring the difference in millimeter between prespecified points
  1-full face 2-subnasal 3-labrale superioris 4- labrale inferioris 5-pogonion 6- corners of the mouth Then the degree of accuracy will be measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmed Farid, Professor of OMFS, Study Director — Cairo University; Sameh Tarek Mekhemar, Head of Department, Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF